CLINICAL TRIAL: NCT01001962
Title: Double Blind Comparison Study of JARDIANCE® (Empagliflozin) in Prehypertensives Type II Diabetics With Metformin
Brief Title: Double Blind Placebo Study of JARDIANCE® (Empagliflozin) in Prehypertensives Type II Diabetics
Acronym: PREHYPD
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Vasilios Kotsis, Prof. Med, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: PREHYPERTENSION
Record Dates: First submitted 2009-10-26; First posted 2009-10-27 (Estimated); Last update posted 2015-04-07 (Estimated); Status verified 2015-04

CONDITIONS: Hypertension; Type II Diabetes
Keywords: Hypertension in type II diabetes; Cardiovascular morbidity and mortality
MeSH Terms: conditions — Hypertension; Diabetes Mellitus, Type 2 | interventions — empagliflozin; Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Metformin (Active Comparator): 527 Patients treated with Metformin 850x2mg titrated to 1000x2mg Daily oral
  Interventions: Drug: Metformin
- Empagliflozin (Active Comparator): 527 Patients treated with empagliflozin 10mg titrated to 25 mg Daily oral
  Interventions: Drug: empagliflozin

INTERVENTIONS:
Drug: empagliflozin — ACTIVE TREATMENT FOR DIABETES
  Other Names: JARDIANCE
  Arms: Empagliflozin
Drug: Metformin — ACTIVE TREATMENT FOR DIABETES
  Other Names: GLUCOPHAGE
  Arms: Metformin

SUMMARY:
Objectives:

Primary

1. Primary prevention of new onset of hypertension

Secondary

1. Reduction of 24h BP in type II diabetics with prehypertension
2. Reduction of non dipping status, day and nighttime BP, morning BP surge in subjects receiving EMPAGLIFLOZIN
3. Reduction in the total cardiovascular risk
4. 3 years morbidity and mortality rates
5. Arterial de-stiffening, reduction in central aortic blood pressure in subjects receiving EMPAGLIFLOZIN

DETAILED DESCRIPTION:
Study rationale: The majority of patients with diabetes are having higher blood pressure than optimal. More than 30% of patients with type II diabetes are prehypertensives with systolic blood pressure between 130 and 140 mmHg. If a drug for diabetes has an impact on blood pressure in such patients then this drug will reduce cardiovascular risk beyond the reduction on glucose levels. There are some evidence that EMPAGLIFLOZIN is reducing blood pressure levels but a comprehensive study is not available.

Timelines and Study duration:

Start date : 01-01-2016 End date : 01-01-2019 Clinical Study Report date: June 2018 Publication date: 2018, 2018, 2019,2020

Methodology:

Inclusion criteria

1. Age between 45 and 60 years.
2. All patients are going to give their informed consent to participate in the study.
3. Patients who are not receiving antihypertensive or diabetes treatment (newly diagnosed diabetics)
4. BP between 130 to 140 mmHg for systolic BP (prehypertensives)
5. Type II diabetes (HbA1c 7.0-8.0)

Exclusion criteria Known oversensitiveness, chronic renal disease (GFR<60 ml/min) or ESRD, heart or respiratory failure, recent MI, shock and pregnancy or lactation.

Study drugs:

Clinical examination 0,1,6,12,24,36 months.

* Duration and follow-up: 3 years
* Collected data: Ambulatory blood pressure monitoring, 24h SBP and DBP in time 0,12, 24 months.
* BMI, waist/hip ratio in time 0, 12, 24,36 months.
* HbA1c, insulin in time 0, 1, 6,12, 24,36 months.
* K, Na, Cr, BUN, Chol, Tg, HDL, LDL,ALT, AST in time 0, 1, 6,12, 24,36 months.

Number of patients: 1054

Sample size justification:

The reduction in mean 24h SBP expected to be 2.5 mmHg. Previous studies from our group reported an 12-14mmHg SD for 24h mean SBP. The sample size required at the two sided 5% significance level and 90% power is 527 patients per drug arm.

Statistics/Data Analysis Stata Estimated sample size for two-sample comparison of means Test Ho: m1 = m2, where m1 is the mean in population 1 and m2 is the mean in population 2

Assumptions:

alpha = 0.0500 (two-sided) power = 0.9000 m1 = 130 m2 = 132.5 sd1 = 12 sd2 = 13 n2/n1 = 1.00

Estimated required sample sizes:

n1 = 527 n2 = 527

Population: Diabetes, prehypertension, outpatients. I

ELIGIBILITY:
Inclusion criteria

1. Age between 45 and 65 years.
2. All patients are going to give their informed consent to participate in the study.
3. Patients who are not receiving antihypertensive or diabetes treatment (newly diagnosed diabetics)
4. BP between 130 to 140 mmHg for systolic BP (prehypertensives)
5. Type II diabetes (HbA1c 7.0-8.0)

Exclusion criteria

1. Known oversensitiveness
2. chronic renal disease (GFR<60 ml/min) or ESRD
3. heart or respiratory failure, recent MI, shock
4. pregnancy or lactation.

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1054 (Estimated)
Dates: Start 2016-01; Primary Completion 2019-01 (Estimated); Study Completion 2020-01 (Estimated)

PRIMARY OUTCOMES:
New onset of hypertension | 36 months

SECONDARY OUTCOMES:
24h blood pressure levels | 36 months
Total cardiovascular risk | 36 months
Morbidity cardiovascular | 36 months
Arterial stiffness | 36 months
Central aortic blood pressure | 36 months
Mortality cardiovascular | 36 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hypertension 24h ABPM center Papageorgiou Hospital, Thessaloniki, Greece

REFERENCES:
- [Derived] Gnesin F, Thuesen ACB, Kahler LKA, Madsbad S, Hemmingsen B. Metformin monotherapy for adults with type 2 diabetes mellitus. Cochrane Database Syst Rev. 2020 Jun 5;6(6):CD012906. doi: 10.1002/14651858.CD012906.pub2. PMID 32501595